CLINICAL TRIAL: NCT00256490
Title: Early Evaluation of the Response of Large B Cell Non Hodgkin's Lymphoma to Chemotherapy by Positron Emission Tomography Coupled With Computed Tomography (PET/CT)
Brief Title: Early Evaluation of the Response of Large B Cell Non Hodgkin's Lymphoma to Chemotherapy by PET/CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eric Turcotte (Other)
Responsible Party: Sponsor-Investigator, Eric Turcotte, MD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRC 05-020; CIMF 2005-01
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Lymphoma, Large-Cell
Keywords: Diffuse large B cells lymphoma; PET/CT; FDG
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

INTERVENTIONS:
Procedure: PET/CT 20 days after the first cycle of chemotherapy

SUMMARY:
Patients affected with non-Hodgkin's large B-cell lymphoma are treated by chemotherapy. The evaluation of the response to this treatment is made by Positron Emission Tomography (PET/CT) in many centres where this technology is available. Presently PET scans and CT scans are being performed before treatment, after 4 cycles of chemotherapy and a few months after the end of treatment.

The goal of this study is to determine if it is possible to evaluate the efficiency of chemotherapy treatments after one cycle of treatment instead of waiting after 4 cycles, using a new scanner that combines PET and CT modalities. Data available from studies on these combined exams suggest that PET/CT helps to rapidly evaluate the response of the chemotherapy treatment. We also want to verify if some pathological characteristics measured from tumor cells will enable doctors to predict in advance the response to treatment.

DETAILED DESCRIPTION:
Participation in this study involves 4 PET/CT exams, which occur before the treatments start, after the first cycle of chemotherapy, after 4 cycles of chemotherapy and then 12 weeks after the end of the treatments. The only additional test performed in this study compared to the regular follow-up of patients that are not in this study is the PET/CT exam after the first cycle. Your participation in this study will not affect treatment since the results of the first PET/CT test will not be communicated. All other tests results will be available in the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed large B cells non Hodgkin's lymphoma, CD20 positive
* Chemotherapy treatments planned (R-CHOP) but not started

Exclusion Criteria:

* Pregnancy (determined by urinary β-HCG and blood test)
* Patients younger than 18 years
* Unable to tolerate the procedure (30 minutes laying down on the back)
* No chemotherapy treatment planned secondary to the patient's health performance
* Previous lymphoma that has been treated with chemotherapy with the exception of stade I lymphoma treated only with radiotherapy.
* All lymphoma other than large cell Non Hodgkin's lymphoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2005-11 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2009-12-01 (Actual)

PRIMARY OUTCOMES:
Disease free survival at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Turcotte, MD, FRCPC, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke; Francois Bénard, MD, FRCPC, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke; Virginie Bruneau, MD, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada